CLINICAL TRIAL: NCT04983953
Title: An Open Label, Single-Center and Random-Selection Retrospective Pivotal Study of Clinical Decision Support System for Intracranial Hemorrhage Using Brain CT Images
Brief Title: Evaluation of Clinical Decision Support System for Intracranial Hemorrhage Using Brain CT Images
Status: Completed | Type: Observational
Sponsor: Heuron Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HR-cHS-01
Record Dates: First submitted 2021-07-29; First posted 2021-07-30 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Intracranial Hemorrhages
MeSH Terms: conditions — Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Abnormal: A patient diagnosed with intracranial haemorrhage after a brain CT scan
  Interventions: Device: cHS
- Normal: A normal person or a patient not diagnosed with intracranial haemorrhage after a brain CT scan
  Interventions: Device: cHS

INTERVENTIONS:
Device: cHS — Clinical decision support system for diagnosing intracranial haemorrhage

SUMMARY:
cHS is a software that has been pre-learned based on a intracranial haemorrhage diagnosis model using brain CT images, and clinical decision support system for diagnosing intracranial haemorrhage by automatically analyzing brain CT images by assisting the medical team.

The specific aims of this study are to evaluate efficacy of cHS for intracranial haemorrhage compared to the sensitivity and specificity levels of predicate device which is currently approved to triage intracranial haemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 19 years old
* Brain CT acquired
* Abnormal cohort: A patient diagnosed with intracranial haemorrhage after a brain CT scan
* Normal cohort: A normal person or a patient not diagnosed with intracranial haemorrhage after a brain CT scan

Exclusion Criteria:

* Patients with brain tumor or cerebral toxoplasmosis
* Patients with brain abscess or brain calcification
* Poor or incomplete brain CT image quality

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (1) Adults over 19 years old (2) Brain CT images acquired (3) who confirmed with intracranial haemorrhage(abnormal cohort) or not intracranial haemorrhage or normal(normal cohort)
Sampling Method: Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of cHS | Within 4 weeks after collecting data
  Sensitivity and specificity of cHS in diagnosis of intracranial haemorrhage based on golden standards

CONTACTS AND LOCATIONS:
Locations (1):
- Gachon University Gil Medical Center, Incheon, Namdong-gu, South Korea

IPD SHARING:
Plan to Share IPD: No